CLINICAL TRIAL: NCT06530693
Title: Optimizing the Prehospital Use of Stroke Systems of Care-Reacting to Changing Paradigms-Implementation (OPUS-i)
Acronym: OPUS-i
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 30716
Record Dates: First submitted 2024-07-03; First posted 2024-07-31 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard transport protocol (Active Comparator): Standard EMS stroke transport protocol
  Interventions: Other: OPUS-i algorithm
- OPUS-i Protocol (Active Comparator): Experimental OPUS-i protocol
  Interventions: Other: OPUS-i algorithm

INTERVENTIONS:
Other: OPUS-i algorithm — A novel pre-hospital algorithm.

SUMMARY:
This interventional trial will compare a novel prehospital stroke transport algorithm (OPUS-i) to a traditional prehospital stroke transport algorithm to improve outcomes in rural stroke patients by determining the effect of implementing a data-driven prehospital stroke algorithm on time to and endovascular therapy. The study consists of a multicenter cohort and will last 24 months but individual subject study duration is 90 days.

DETAILED DESCRIPTION:
Stroke is the fifth leading cause of death in the United States (U.S.) and causes one in six deaths from cardiovascular disease. Intravenous thrombolysis (IVT), unless contraindicated, is the standard of care for acute ischemic strokes (AIS) presenting within 4.5 hours of last known well. IVT plus endovascular therapy (EVT) is standard of care for the typically debilitating large vessel occlusion strokes (LVOS), which represent 30% of AIS. However, only a limited number of stroke centers provide EVT. Currently only 12% of all stroke patients are treated with IVT and only 8% of patients are treated with EVT. Therefore, optimizing prehospital systems of care to provide timely IVT and EVT to all patients.

Most stroke patients arrive at the hospital by Emergency Medical Services (EMS). EMS clinicians use various stroke assessment tools to triage patients to the appropriate level of stroke center. Unfortunately, these prehospital stroke screen tools are imprecise and can delay care for LVOS patients. The choice of transport destination may vary by geography. In an urban area, where several stroke centers of varying capability may be concentrated in a small geographical area, there is negligible impact to the healthcare system if an ambulance bypasses the closest hospital for an ESC. In a more rural area, the decision regarding hospital transport destinations has greater implications. Transporting a patient to a farther ESC will result in a longer transport time and take an ambulance out of its primary coverage for a prolonged time. However, transporting rural stroke patients to their local non-ESC may worsen their clinical outcomes by delaying the time to EVT.

Therefore, we propose to implement the novel OPUS-i prehospital stroke transport algorithm to improve outcomes for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical impression of stroke/TIA by EMS clinicians

Exclusion Criteria:

* Age < 18 years
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Time from stroke onset to endovascular therapy | From time of stroke onset to endovascular therapy, assessed on day 0 of admission
  This outcome will assess process measures for acute stroke patients

SECONDARY OUTCOMES:
Time from stroke onset IVT | From time of stroke onset to IVT, Assessed on day 0 of admission
  This outcome will assess process measures for acute stroke patients
Rate of bypass of non-ESCs for rural and urban patients. | The percentage of patients bypassed from non-ESCs to ESCs, assessed on day 0 of admission
  This outcome will assess rates of bypass to narrow the disparity between urban and rural patients.
Rate of bypass of non-ESCs for rural and urban patients. | Modified Rankin Scale of 0-2 at 90 days in patients for all stroke patients.
  This outcome will assess good functional outcomes after stroke.
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in LVOS | Modified Rankin Scale of 0-2 at 90 days in patients with large vessel occlusion stroke.
  This outcome will assess good functional outcomes after stroke for the subgroup of LVOS patients
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in patients with LVOS | Modified Rankin Scale of 0-2 at 90 days for patients with intracranial hemorrhage
  This outcome will assess good functional outcomes in patients with ICH.
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in patients with non-LVO AIS | Modified Rankin Scale of 0-2 at 90 days for patients with non-LVO AIS
  This outcome will assess good functional outcomes in patients with non-LVO AIS
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes. | Modified Rankin Scale of 0-1 at 90 days for all patients.
  This outcome will assess excellent functional outcome after stroke.
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in LVOS | Modified Rankin Scale of 0-1 at 90 days in patients with LVOS.
  This outcome will assess excellent functional outcomes after stroke in patients with LVOS
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in ICH. | Modified Rankin Scale of 0-1 at 90 days for patients with intracranial hemorrhage.
  This outcome will assess excellent functional outcomes after ICH.
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in non-LVO AIS. | Modified Rankin Scale of 0-1 at 90 days for patients with non-LVO AIS
  This outcome will assess excellent functional outcomes after non-LVO AIS.
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes | up to 90 days
  This will assess good functional outcomes after stroke.
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in LVOS | up to 90 days
  This outcome will assess good functional outcomes after stroke for the subgroup of LVOS patients
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in patients with LVOS | up to 90 days
  This outcome will assess good functional outcomes in patients with ICH.
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in patients with non-LVO AIS | up to 90 days
  This outcome will assess good functional outcomes in patients with non-LVO AIS
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes. | up to 90 days
  This outcome will assess excellent functional outcome after stroke.
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in LVOS. | up to 90 days
  This outcome will assess excellent functional outcomes after stroke in patients with LVOS.
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in ICH | up to 90 days
  This outcome will assess excellent functional outcomes after ICH.
To evaluate the effect of a novel prehospital stroke transport algorithm on stroke outcomes in non-LVO AIS | up to 90 days
  This outcome will assess excellent functional outcomes after non-LVO AIS.
To evaluate the effect of a novel prehospital stroke transport algorithm on patients with hyperacute strokes To evaluate the effect of a novel prehospital stroke transport algorithm on patients with hyperacute strokes | Modified Rankin Scale of 0-2 at 90 days in patients with last known well to hospital arrival of <4 hour
  This outcome will assess good functional outcomes after hyperacute ischemic stroke.
To evaluate the effect of a novel prehospital stroke transport algorithm on all-cause mortality | All-cause mortality at 90 days
  This outcome will assess all-cause mortality at 90 days.
To evaluate the effect of a novel prehospital stroke transport algorithm on all-cause mortality in LVOS patients | All-cause mortality at 90 days for LVOS patients
  This outcome will assess all-cause mortality at 90 days for LVOS patients.
To evaluate the effect of a novel prehospital stroke transport algorithm on all-cause mortality in patients with ICH | All-cause mortality at 90 days for patients with ICH
  This outcome will assess all-cause mortality at 90 days for patients with ICH.
To evaluate the effect of a novel prehospital stroke transport algorithm on all-cause mortality for patients with non-LVO AIS | All-cause mortality at 90 days for patients with non-LVO AIS
  This outcome will assess all-cause mortality at 90 days for patients with non-LVO AIS.
To evaluate process measures in stroke care | up to 90 days
  This outcome will assess the effect of the OPUS-i algorithm on time from stroke onset to IVT
To evaluate process measures in stroke care | up to 90 days
  This outcome will assess the effect of the OPUS-i algorithm on time from stroke onset to EVT
To evaluate process measures in stroke care | up to 90 days
  Rate of IVT
To evaluate process measures in stroke care | up to 90 days
  Rate of EVT
To compare the above processes and outcomes in rural versus urban patients | up to 90 days
  mRS in rural vs urban patients

CONTACTS AND LOCATIONS:
Overall Officials: Derek Isenberg, MD, Principal Investigator — Lewis Katz School of Medicine at Temple University
Locations (1):
- 3401 N Broad street, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year after study completion